CLINICAL TRIAL: NCT03098433
Title: Effects of Liothyronine on Energy Expenditure and Cardiovascular Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HM20005777
Record Dates: First submitted 2017-03-07; First posted 2017-03-31 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Triiodothyronine; Thyroxine

STUDY DESIGN:
Intervention Model Description: double blind, crossover
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Liothyronine (Experimental): Each participant will receive a single dose of lithyronine
  Interventions: Drug: Liothyronine
- Levothyroxine (Active Comparator): Each participant will receive a single dose of levothyroxine
  Interventions: Drug: Levothyroxine
- Placebo (Placebo Comparator): Each participant will receive a single dose of placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Liothyronine — Single dose
  Arms: Liothyronine
Drug: Levothyroxine — Active comparator
  Arms: Levothyroxine
Drug: Placebos — Placebo
  Arms: Placebo

SUMMARY:
This study will assess the short term effects of a single dose of liothyronine on the cardiovascular system and energy expenditure

ELIGIBILITY:
Inclusion Criteria:

* BMI >20<30 kg/m2
* TSH >0.5<5.0 mcIU/mL
* Negative TPO antibodies

Exclusion Criteria:

* Pregnancy
* Use of prescription drugs
* Diabetes mellitus
* Coronary artery disease
* Hypertension
* Anemia
* Renal insufficiency
* Liver disease or ALT >2.5 x the upper laboratory reference limit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco S Celi, MD, MHSc., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen S, Wohlford GF, Vecchie' A, Carbone S, Yavuz S, Van Tassell B, Abbate A, Celi FS. Acute Effects of Liothyronine Administration on Cardiovascular System and Energy Metabolism in Healthy Volunteers. Front Endocrinol (Lausanne). 2022 Feb 28;13:843539. doi: 10.3389/fendo.2022.843539. eCollection 2022. PMID 35295986

RESULTS

PARTICIPANT FLOW:
Groups:
- Three Treatments in Random Order: Each participant will receive a single dose of lithyronine, a single dose of levothyroxine, and a single dose of placebo, in a random order.
  Information on the order of treatments was not collected.
  Participants will attend three study visits. At the first study visit one of the three treatments will be randomly selected and administered.
  At the second study visit one of the remaining two treatments will be randomly selected and administered.
  At the third study visit the final treatment will be administered.
  The order of administration will not be analyzed therefore all participants are part of a single arm.
Period: Overall Study
Arm/Group | Three Treatments in Random Order
Started | 22
Completed | 12
Not Completed | 10
Not completed — Withdrawal by Subject | 10

BASELINE CHARACTERISTICS:
Groups:
- Three Treatments in Random Order: Each participant will receive a single dose of lithyronine, a single dose of levothyroxine, and a single dose of placebo, in a random order.
  Information on the order of treatments was not collected.
  Participants will attend three study visits. At the first study visit one of the three treatments will be randomly selected and administered.
  At the second study visit one of the remaining two treatments will be randomly selected and administered.
  At the third study visit the final treatment will be administered.
  The order of administration will not be tracked.
Arm/Group | Three Treatments in Random Order
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Output
Description: Cardiac output measured by Echocaridogram, Difference in Stroke Volume Pre- and Post- Drug Administration
Time Frame: five hours
Population: I participant did not undergo echocardiogram
Measure: Mean (Standard Deviation); unit: millilitres
Groups:
- Three Treatments in Random Order: Each participant will receive a single dose of lithyronine, a single dose of levothyroxine, and a single dose of placebo, in a random order
  Information on the order of treatments was not collected.
  Participants will attend three study visits. At the first study visit one of the three treatments will be randomly selected and administered.
  At the second study visit one of the remaining two treatments will be randomly selected and administered.
  At the third study visit the final treatment will be administered.
  The order of administration will not be tracked.
Arm/Group | Three Treatments in Random Order
Number analyzed (Participants) | 11
millilitres
  Liothyronine | -3.7 (8.8)
  Levothyroxine | -1.4 (6.5)
  Placebo | 1 (6.2)

2. Secondary Outcome: Energy Expenditure
Description: Energy expenditure measured by Whole-Room Indirect Calorimeter, Difference in energy Expenditure Pre- and Post- Drug Administration Kcal
Time Frame: five hours
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Three Treatments in Random Order
Number analyzed (Participants) | 12
kcal
  Liothyronine | 0.006 (0.067)
  Levothyroxine | -0.05 (0.058)
  Placebo | -0.007 (0.062)

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Three Treatments in Random Order
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT03098433/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03098433/Prot_SAP_002.pdf